CLINICAL TRIAL: NCT04962490
Title: Study of the Repair of Flexor Tendons of the Hand: Epidemiological and Prognostic Factors Associated With Tendon Injuries in Zone II
Brief Title: Study of the Repair of Flexor Tendons of the Hand
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TFM-2021-34
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-03

CONDITIONS: Tendon Injury - Hand
Keywords: tendon, flexor, hand
MeSH Terms: interventions — Replantation; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Repair: suture, reinsertion, tendon graft, surgery in two stages (Hunter, Paneva Holevich) — Repair tendon flexor sections in the hand: Suture, reinsertion, tendon graft, surgery in two stages (Hunter, Paneva Holevich). The surgery depends on the anatomical area of the tendon section and the time between the injury and the operation.

SUMMARY:
Injury to the flexor tendons of the fingers of the hand is a frequent and disabling injury, since it produces tendon retraction and functional limitation. A prompt and adequate diagnosis and treatment is required to minimize the risk of tendon retraction, re-rupture, reoperation rate, and the presence of tendon adhesions that limit the range of motion. On occasions, the limitation of the articular balance of the MCP, PIP and DIP joints generates a loss of strength and difficult in completely closing the fingers to the palm of the hand.

DETAILED DESCRIPTION:
To retrospectively evaluate the results obtained with the suture/ reinsertion of the flexor tendons of the hand, in the acute, subacute and chronic phases, treated surgically in our center between the years 2000 and 2021.

To evaluate the clinical and functional results obtained in patients who underwent surgery for a section of the flexor tendons, superficial, profundus or both, preferably in zone II of the hand. The investigators evaluate the epidemiological and prognostic factors associated with the injury, in the different phases and anatomical zones.

The researchers evaluate the functional results:

Pain at rest with movements: Assessed using the visual analogue pain scale (VAS Scale from 0 to 10).

Joint balance / Range of motion of the MCP, PIP, DIP joints. Evaluation by digital goniometer. Evaluation using Buck-Gramcko (1976) and using the Tang (2007) criteria.

Grip strength. Evaluation using a Jamar dynamometer. Functional rating scales: QuickDASH Score Reoperation rate: 1) For re-rupture / re-suture, 2) For infection, 3) For excision of tendon adhesions: arthrolysis and tendolysis, 4) For tendon transfer 5) For tendon graft placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with section of the superficial and / or profundus flexor tendons in the hand.
* Patients with section of the flexor tendon in the thumb
* Tendon injury in any anatomical area
* In the acute, subacute or chronic phases of the disease
* Associated or not with fractures
* Associated or not with arterial or nerve injuries

Exclusion Criteria:

* Previous bone disease
* History of tendon injury to the extensor or flexor tendons
* Joint stiffness prior to tendon section
* Rheumatic arthropathy
* History of operations in the same area.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients between 18 and 85 years of age who have suffered a hand injury with section / s of the superficial and / or profundus flexor tendons, or both in hand; and flexor tendon in the thumb.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Range of motion (ROM) | 12 months
  Change in the mobility of the MCP, PIP and DIP joints. Evaluation with goniometer (cm)
Grip Strength | 12 months
  Change of strength with respect to the contralateral hand. Evaluation with Jamar Dinamometer (Kg)
Chronic residual pain | 12 months
  Evaluation residual pain at rest and with activity with the Visual Analogue Scale (values from 0 to 10; 0 is the better outcome and 10 is the worse outcome).

SECONDARY OUTCOMES:
Epidemiological variables age, sex, smoker, diabetes, heart disease, other diseases (lung, kidney, etc.). | 12 months
  Evaluacion of epidemiological factors associated with outcomes in flexor injuries.
Trauma variables | 12 months
  Affected finger, dominant hand, involvement of one or more fingers, type of injury (complete / partial section / association with fractures /association with arterial injury/ association with nerve injury/ section only FP or section FS plus FP).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, MD, Ph D, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Claudia Erika Delgado Espinoza, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Doyle JR. Anatomy of the flexor tendon sheath and pulley system: a current review. J Hand Surg Am. 1989 Mar;14(2 Pt 2):349-51. doi: 10.1016/0363-5023(89)90110-x. PMID 2732428
- [Result] Manske PR. Flexor tendon healing. J Hand Surg Br. 1988 Aug;13(3):237-45. doi: 10.1016/0266-7681_88_90077-0. PMID 3049854
- [Result] Tang JB. Indications, methods, postoperative motion and outcome evaluation of primary flexor tendon repairs in Zone 2. J Hand Surg Eur Vol. 2007 Apr;32(2):118-29. doi: 10.1016/J.JHSB.2006.12.009. Epub 2007 Feb 12. PMID 17298858
- [Result] Tang JB. Flexor tendon repair in zone 2C. J Hand Surg Br. 1994 Feb;19(1):72-5. doi: 10.1016/0266-7681(94)90054-x. PMID 8169485
- [Result] Moriya K, Yoshizu T, Tsubokawa N, Narisawa H, Matsuzawa S, Maki Y. Outcomes of flexor tendon repairs in zone 2 subzones with early active mobilization. J Hand Surg Eur Vol. 2017 Nov;42(9):896-902. doi: 10.1177/1753193417715213. Epub 2017 Jun 13. PMID 28610452
- [Result] Amadio PC, Hunter JM, Jaeger SH, Wehbe MA, Schneider LH. The effect of vincular injury on the results of flexor tendon surgery in zone 2. J Hand Surg Am. 1985 Sep;10(5):626-32. doi: 10.1016/s0363-5023(85)80197-0. PMID 4045137
- [Result] Lundborg G, Myrhage R, Rydevik B. The vascularization of human flexor tendons within the digital synovial sheath region--structureal and functional aspects. J Hand Surg Am. 1977 Nov;2(6):417-27. doi: 10.1016/s0363-5023(77)80022-1. PMID 925330
- [Result] Buck-Gramcko D, Dietrich FE, Gogge S. [Evaluation criteria in follow-up studies of flexor tendon therapy]. Handchirurgie. 1976;8(2):65-9. German. PMID 992488
- [Result] Tang JB. Outcomes and evaluation of flexor tendon repair. Hand Clin. 2013 May;29(2):251-9. doi: 10.1016/j.hcl.2013.02.007. PMID 23660061
- [Result] Strickland JW. Development of flexor tendon surgery: twenty-five years of progress. J Hand Surg Am. 2000 Mar;25(2):214-35. doi: 10.1053/jhsu.2000.jhsu25a0214. No abstract available. PMID 10722813